CLINICAL TRIAL: NCT06284070
Title: Application of FAPI and FDG PET Imaging in Patients With Different Types of Cancer
Status: Recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Xiao Chen, Director of Nuclear Medicine Department, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: 202433
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cancer
Keywords: FAPI; cancer; FDG; PET
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer associated fibroblasts (CAFs) can promote tumor cell proliferation, migration, invasion, and angiogenesis through immunosuppressive effects and the production of mediators, thereby promoting tumor growth and progression. The characteristic of CAFs is high expression of fibroblast activation protein (FAP). In approximately 90% of epithelial derived tumors, FAP is highly overexpressed on the membrane of CAFs. Contrary to CAFs, FAP expression is lower or absent in normal tissues. Therefore, FAP inhibitors (FAPI) targeting FAP can overcome the limitations of 18F-2-fluoro.2-deoxy-D-glucose fluorodeoxyglucose(18F-FDG) PET imaging. But like 18F-FDG, wound healing, fibrosis, and inflammation can also uptake FAPI.. Therefore, a comparison of the performance of 18F-FDG and 18F-FAPI PET imaging in diagnosing primary and metastatic lesions of various types of cancer is conducted to evaluate the potential value of these new radiopharmaceuticals as effective alternatives to 18F-FDG, highlighting their advantages and limitations.

DETAILED DESCRIPTION:
This study is a prospective, single study and has been approved by the ethics committee. The subjects of this studywere from January 1,2024 to December 31, 2029.The detailed description is as follows:

1. Patients: The subjects we selected are adults who are not restricted by gender. For details, please refer to the "Eligibility Criteria" column.
2. Clinical data collection: Record the course of disease, laboratory tests (tumor markers, inflammatory markers), PET examinations, and follow-up related imaging (ultrasound, CT, or magnetic resonance imaging（MRI）) information of all patients.
3. CT or MRI image analysis: Record the location and number of lesions, measure the long diameter of the primary and metastatic lesions, and the short diameter of lymph nodes on CT or MRI images.
4. PET image analysis: Record and evaluate the following indicators: the maximum, mean and peak standardized uptakevalue (SUVmax, SUVmean and SUVpeak), Metabolic lesion volume (MLV), total lesion glycolysis (TLG).
5. Statistical analysis: Use descriptive statistical methods to compare the age of patients and the standardized uptake values of FDG and FAPI. Normal distribution data is represented as mean ± standard deviation, while non normal distribution data is represented as median with IQR. Compare the normal distribution data between two groups using paired two sample t-test, and compare the non normal distribution data between two groups using McNemar test. Using a four grid table McNemar χ Compare the diagnostic efficacy of 18F-FDG PET and 18F-FAPI PET through 2 tests, calculate and compare the sensitivity, specificity, positive predictive value, negative predictive value, and accuracy of 18F-FDG and 18F-FAPI PET. Due to the potential impact of tumor type on diagnosis, subgroup analysis was conducted on the diagnostic efficacy of 18F-FDG PET and 18F-FAPI PET. Due to the possibility of multiple metastatic lesions in a given participant, the diagnostic results may be correlated within the participant. Therefore, sensitivity analysis of metastatic lesions is also performed based on a generalized linear mixed effects model by combining this correlation between different lesions within the same participant. Double tailed P<0.05 indicates a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years old);
2. Suspected or newly diagnosed malignant tumor patients;
3. Patients who underwent 18F-FDG and 18F-FAPI PET scans within one week;
4. Patients who are able to provide informed consent forms (signed by participants, parents, or legal representatives) and consent forms in accordance with the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

1. Pregnant women;
2. Scanned images with poor image quality due to factors such as body movement;
3. Patients with mental illness or other unsuitable conditions for examination, poor compliance, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects we selected are adults who are not restricted by gender. For details, please refer to the "EligibilityCriteria" colymn.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | Completed within half year after end of the study
  The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 18F-FDG and 18F-FAPI PET were calculated and compared to evaluate the diagnostic efficacy.

SECONDARY OUTCOMES:
SUV | Completed within one week after PET examination
  Standardized uptake value (SUV) of 18F-FDG and 18F-FAPI for each target lesion of subject or suspected primary tumor or/and metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, Daping Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hirmas N, Hamacher R, Sraieb M, Kessler L, Pabst KM, Barbato F, Lanzafame H, Kasper S, Nader M, Kesch C, von Tresckow B, Hautzel H, Aigner C, Glas M, Stuschke M, Kummel S, Harter P, Lugnier C, Uhl W, Hadaschik B, Grunwald V, Siveke JT, Herrmann K, Fendler WP. Diagnostic Accuracy of 68Ga-FAPI Versus 18F-FDG PET in Patients with Various Malignancies. J Nucl Med. 2024 Mar 1;65(3):372-378. doi: 10.2967/jnumed.123.266652. Epub 2024 Feb 8. PMID 38331453
- See also: Diagnostic Accuracy of 68Ga-FAPI Versus 18F-FDG PET in Patients with Various Malignancies — https://pubmed.ncbi.nlm.nih.gov/38331453/